CLINICAL TRIAL: NCT04620057
Title: Effects of Oral Supplementation of Butyrate in Children With Obesity
Brief Title: Effects of Butyrate Against Pediatric Obesity
Acronym: BAPO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Roberto Berni Canani, MD, PhD, Chief of the Pediatric Allergy Program at the Department of Translational Medical Science Chief of the ImmunoNutritionLab at CEINGE - Advanced Biotechnologies, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 29ES20
Record Dates: First submitted 2020-10-26; First posted 2020-11-06 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity | interventions — Butyrates

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Butyrate + standard care for pediatric obesity (Experimental): standard care for pediatric obesity + sodium butyrate (20 mg/kg body weight/day)
  Interventions: Dietary Supplement: butyrate
- placebo + standard care for pediatric obesity (Placebo Comparator): standard care for pediatric obesity + placebo (cornstarch)
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: butyrate — sodium butyrate (20 mg/kg body weight/day)
  Arms: Butyrate + standard care for pediatric obesity
Other: placebo — cornstarch
  Arms: placebo + standard care for pediatric obesity

SUMMARY:
Worldwide obesity is a public health concern that is defined by the World Health Organization as abnormal or excessive fat accumulation that may impair health. The main drivers of obesity pathogenesis seem to be a long-term of energy discrepancy between too many calories consumed and an increase of sedentary behavior. A growing body of evidence suggests that the set of microbes that live within the digestive tract, making up the gut microbiota (GM), play a metabolic role in energy regulation and substrate metabolism. Various factors can impact GM, one of these are dietary compounds that deeply affect the growth and metabolism of gut bacteria, since fermentation of nutrients is one core function of the intestinal microbes. Among fermentation products an array of small organic metabolites are short-chain fatty acids (SCFAs) acetate, propionate and butyrate. Among SCFAs, the C-4 fatty acid butyrate, the main fuel for the colonocytes, might have a potential in alleviating obesity and related metabolic complications. Butyrate could act as a regulator of body weight: a reasonable speculation is that butyrate acts on components of the energy balance, promoting energy expenditure and/or reducing energy intake. Preclinical studies have shown that butyrate supplementation prevent high-fat diet-induced obesity and it is able to treat obesity. With the sharp increase of obesity prevalence seen in the pediatric population, novel insights are necessary to counteract this epidemic disease, the outcome of the study is to see whether oral butyrate supplementation could exert similar effect in obese children.

ELIGIBILITY:
Inclusion Criteria:

* Children/adolescents with diagnosis of obesity (BMI >95° percentile for age and sex) observed at Pediatric Section of Department of Translational Medical Sciences (University of Naples Federico II)

Exclusion Criteria

* Age at enrollment <5 or >17 years
* BMI <95° percentile for age and sex
* Patients under pharmacological treatment for obesity (metformin)
* Patients assuming vitamin E,
* Patients assuming pre-, pro- or synbiotics
* Simultaneous presence of other chronic diseases unrelated to obesity:

  * cancer,
  * immunodeficiency,
  * cystic fibrosis,
  * allergies,
  * celiac disease,
  * autoimmune diseases,
  * neuropsychiatric disorders,
  * type 1 diabetes,
  * inflammatory bowel diseases,
  * malformations of urinary or gastrointestinal or respiratory tract,
  * chronic lung diseases, genetic and metabolic diseases,
  * chronic hematological diseases.
* History of surgery for the treatment of obesity
* Any medical condition that may interfere with participation in this study
* Participation in other clinical trials still in progress

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
BMI z-score change | after 6 months from the start of intervention
  BMI z-score change at least of ≥ 0.25

SECONDARY OUTCOMES:
waist circumference | after 6 months from the start of intervention
  mean waist circumference change
HOMA index change | after 6 months from the start of intervention
  mean of HOMA index change
fasting glucose change | after 6 months from the start of intervention
  mean of fasting glucose change
fasting insulin change | after 6 months from the start of intervention
  mean of fasting insulin change
total cholesterol change | after 6 months from the start of intervention
  mean of total cholesterol change
Low density Lipoprotein cholesterol change | after 6 months from the start of intervention
  mean of Low density Lipoprotein cholesterol change
High density Lipoprotein cholesterol change | after 6 months from the start of intervention
  mean of high density Lipoprotein cholesterol change
plasma triglycerides change | after 6 months from the start of intervention
  mean of plasma triglycerides change
micro RNA 221- expression | after 6 months from the start of intervention
  mean of mir221- expression
serum ghrelin | after 6 months from the start of intervention
  mean of serum ghrelin
serum Interleukin-6 | after 6 months from the start of intervention
  mean of Interleukin-6
composition of the intestinal microbiota (metagenomics characteristics) | after 6 months from the start of intervention
  evaluation of gut microbiota structure by shotgun analysis

CONTACTS AND LOCATIONS:
Locations (1):
- University of Naples Federico II, Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Coppola S, Nocerino R, Paparo L, Bedogni G, Calignano A, Di Scala C, de Giovanni di Santa Severina AF, De Filippis F, Ercolini D, Berni Canani R. Therapeutic Effects of Butyrate on Pediatric Obesity: A Randomized Clinical Trial. JAMA Netw Open. 2022 Dec 1;5(12):e2244912. doi: 10.1001/jamanetworkopen.2022.44912. PMID 36469320